CLINICAL TRIAL: NCT05725031
Title: Intubation Conditions After Rapid Sequence Induction Using Different Doses of Rocuronium with Ephedrine Pretreatment: a Randomized Controlled Trial
Brief Title: Intubation Conditions After RSI Using Rocuronium with Ephedrine Pretreatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amal Ahmed Eldemohi, Resident of Anesthesiology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Eph-Roc
Record Dates: First submitted 2023-01-25; First posted 2023-02-13 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Rapid Sequence Induction and Intubation
MeSH Terms: interventions — Ephedrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ER6 (Experimental): to receive rocuronium 0.6 mg/kg with ephedrine pretreatment
  Interventions: Drug: Ephedrine; Drug: Rocuronium 0.6
- ER8 (Experimental): to receive rocuronium 0.8 mg/kg with ephedrine pretreatment
  Interventions: Drug: Ephedrine; Drug: Rocuronium 0.8
- R12 (Active Comparator): to receive rocuronium 1.2 mg/kg with no pretreatment
  Interventions: Drug: Rocuronium 1.2

INTERVENTIONS:
Drug: Ephedrine — 70 μg/kg as pretreatment
  Arms: ER6; ER8
Drug: Rocuronium 0.6 — 0.6 mg/kg
  Arms: ER6
Drug: Rocuronium 0.8 — 0.8 mg/kg
  Arms: ER8
Drug: Rocuronium 1.2 — 1.2 mg/kg
  Arms: R12

SUMMARY:
This trial will study if ephedrine pretreatment before low doses of rocuronium (0.6 or 0.8 mg/kg) would provide similar intubating conditions as with the high dose of 1.2 mg/kg in patients undergoing RSII.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II

Exclusion Criteria:

* Neuromuscular disease: myopathies
* On drugs that interact with the neuromuscular junction or ephedrine
* Cardiovascular disease: hypertension or ischemic heart disease
* Increased risk of pulmonary aspiration:

  * GERD
  * Pregnancy
* Anticipated airway difficulties:

  * Mallampati grade III or IV
  * Obesity (BMI ≥30 kg/m2),
* Hypersensitivity to any of the study drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Intubation conditions | after 60 seconds of rocuronium administration
  Evaluation of intubation conditions after rapid sequence induction using rocuronium 0.6 or 0.8 mg/kg with ephedrine pretreatment, compared with 1.2 mg/kg, according to the criteria of the Good Clinical Research Practice (GCRP) in pharmacodynamic studies of NMBAs (Fuchs-Buder et al., 2007), which assess each of the following variables for their qualities described as: (excellent, good, poor)
  * ease of laryngoscopy (easy, fair, difficult)
  * vocal cords position (abducted, intermediate, closed)
  * reaction to tracheal tube insertion and cuff inflation (coughing: none, slight, vigorous)
  The 3 variables will be combined to describe intubation conditions as:
  * Excellent: if all qualities are excellent
  * Good: if all qualities are either excellent or good
  * Poor: if there is a single poor quality

SECONDARY OUTCOMES:
Heart rate | every minute of the first 5 minutes of intubation
  Following up the heart rate on the monitor
Mean arterial pressure | every minute of the first 5 minutes of intubation
  Following up the mean arterial pressure by noninvasive blood pressure monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No